CLINICAL TRIAL: NCT01928277
Title: Weaning From Mechanical Ventilation: Spontaneous Breathing Trial and the Assessment of Work of Breathing
Status: Completed | Type: Observational
Sponsor: University of Tromso (Other)
Collaborators: Nord-Trøndelag University College (Other); Helse Nord-Trøndelag HF (Other)
Responsible Party: Sponsor
Other Study IDs: 2012/1230(REK)
Record Dates: First submitted 2013-06-28; First posted 2013-08-23 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Weaning Failure
Keywords: Symptom assessment agreement; Work of breathing

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ICU-patients: ICU-patients weaning form mechanical ventilation

SUMMARY:
The main objective of the study is to examine the extent of agreement between patient and health care provider assessments of work of breathing and the association of agreement with demographic- and disease-related factors.

DETAILED DESCRIPTION:
Mechanical ventilation is among the most common interventions in the intensive care unit (ICU). Over the last two decades, numerous studies have investigated methods to improve outcomes of patients receiving mechanical ventilation. Despite this proliferation of data, a large, multi-national cohort study found clinical outcomes such as duration of ventilation and ICU stay have not improved significantly between1998 to 2004.

It is recommended that weaning should be considered as early as possible in the patient trajectory and spontaneous breathing trials (SBT) attempted, as SBT are the best diagnostic criteria to determine extubation readiness. The decision of ready to extubate is considered complex because both delayed and failed extubations are associated with increased ventilator time and increased mortality. It is shown that dyspnea occurs among nearly half of ventilator patients and is strongly associated with anxiety and delayed extubation. Between 30-75% of ICU patients report anxiety where dyspnea, impaired communication skills, and sleep disturbances may be predisposing factors. The assessments of work of breathing and clinical deterioration are important sub-categories in clinical judgment for determining weaning tolerance.

There is little evidence whether the patients experiences of work of breathing is correlating with physicians and nurses. Hence, we suggest the need to evaluate the interobserver agreement for clinical assessment in weaning.

The main objective of the study is to examine the extent of agreement between patient and health care provider assessments of work of breathing and the association of agreement with demographic- and disease-related factors.

ELIGIBILITY:
Inclusion Criteria:

* Patients using artificial airway (intubation and / or tracheostomy)
* Duration of mechanical ventilation longer than 24 hours
* weaning from mechanical ventilation
* 18 years of age or older
* Motor Activity Assessment Scale (MAAS) 3-4

Exclusion Criteria:

* less than 18 years of age
* insufficient command of the language spoken in the study center
* serious brain damage
* withdrawal of consent at any stage of the research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU-patients weaning from mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
The extent of agreement between patient and provider assessment of work of breathing | 30 minutes
  30 minutes after the initiating of SBT, the patient is asked to rate the sense of work of breathing on a numerous rating scale (NRS, 0-10) At the same time nurse and physician are asked to assess the patients work of breathing on a NRS

SECONDARY OUTCOMES:
The extent of agreement between patient and provider assessment of sense of security | 30 minutes
  30 minutes after the initiating of SBT, the patient is asked to rate the sense of security on a numerous rating scale (NRS, 0-10) At the same time nurse and physician are asked to assess the patients sense of security on a NRS
The extent of agreement between patient and provider assessment of sense of breathing progress | 30 minutes
  30 minutes after the initiating of SBT, the patient is asked to rate the sense of breathing progress on a numerous rating scale (NRS, 0-10) At the same time nurse and physician are asked to assess the patients' breathing progress on a NRS

OTHER OUTCOMES:
Association of agreement of work of breathing with demographic- and disease-related factor (Age, gender, SOFA-score, ventilator time, ICU-mortality) | within the first 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Sissel L Storli, PhD, Principal Investigator — University of Tromso
Locations (2):
- Norway (2):
  - Levanger Hospital, Levanger, Levanger
  - St.Olav Hospital, Trondheim, Trondheim

REFERENCES:
- [Derived] Haugdahl HS, Storli SL, Meland B, Dybwik K, Romild U, Klepstad P. Underestimation of Patient Breathlessness by Nurses and Physicians during a Spontaneous Breathing Trial. Am J Respir Crit Care Med. 2015 Dec 15;192(12):1440-8. doi: 10.1164/rccm.201503-0419OC. PMID 26669474